CLINICAL TRIAL: NCT04868812
Title: Histological Modifications of Postmenopausal Vaginal Mucosa After Repeated CO2 Laser
Brief Title: Histological Modifications of Postmenopausal Vaginal Mucosa After Repeated Carbon Dioxide (CO2) Laser Treatment
Acronym: REPLAMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPLAMOD
Record Dates: First submitted 2020-11-27; First posted 2021-05-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Vaginal Atrophy; Breast Cancer Female; Dyspareunia
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental): All participants will be screened to ensure inclusion/exclusion criteria are met. A biopsy will be taken from each patient one month before the first laser treatment and one month after the last laser treatment. The MonaLisa treatment will be performed monthly for 3 months. A clinical evaluation will be recorded for each patient using validated questionnaires at baseline and one month after the last procedure.
  Interventions: Device: SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy

INTERVENTIONS:
Device: SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy — SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy; MonaLisa Touch CO2 fractionated laser

SUMMARY:
To assess the long-term histological and clinical efficacy of MonaLisa Touch procedure for the management of the Genitourinary Syndrome of Menopause (GSM) in postmenopausal female patients.

DETAILED DESCRIPTION:
The investigator propose a prospective case series of 15 postmenopausal women with bothersome symptoms of GSM treated with MonaLisa Touch CO2 laser. The investigator hypothesize that even in the long term MonaLisa Touch will significantly improve GSM histologically and clinically from baseline.

The primary outcome objective of the study is to evaluate the histological modifications of the vaginal mucosa after repeated CO2 Monalisa Touch laser treatment. The investigator shall evaluate the role of this treatment by calculating the difference in vaginal epithelial thickness between the biopsy obtained before the start of laser treatment and the biopsy obtained after treatment. In addition, the study will analyze the safety of repeated laser treatments verifying the absence of fibrosis formation in the vaginal mucosa. Secondary objectives of the study will include an evaluation of the clinical effects associated with repeated Monalisa Touch CO2 laser treatments using validated questionnaires.

All participants will be screened to ensure inclusion/exclusion criteria are met. A biopsy will be taken from each patient one month before the first laser treatment and one month after the last laser treatment. The MonaLisa treatment will be performed monthly for 3 months. MonaLisa treatment with fractional microablative laser system. For subjects with concomitant vulvar symptoms, vulvar treatment will be done. Biopsy samples will be analyzed with Hematoxylin- Eosin and Trichrome staining, Periodic acid-Schiff (PAS) reaction for glycogen and immunohistochemistry for CD34, a vessel marker. All clinical questionnaires will be assessed at baseline and at one month after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Italian speaking and able to give informed consent.
* Menopausal females with absence of menstruation for at least 12 months.
* Presence of GSM symptoms.
* Completion of at least two cycles of three laser treatments sessions in previous years.
* Prolapse stage < II, according to the pelvic organ prolapse quantification (POP-Q) system.
* No pelvic surgery within 6 months prior to treatment.
* Understanding and acceptance to the obligation to return to all scheduled visits and follow-ups.

Exclusion Criteria:

* Inability of give informed consent
* History of vulvovaginal condyloma, vaginal intraepithelial neoplasia (VAIN), vaginal carcinoma, lichen sclerosis, lichen planus.
* History of cancers of the lower genital tract (cervix, uterus, vagina).
* History of pelvic radiotherapy.
* Personal history of genital fistula, a thin recto-vaginal septum as determined by the investigator or personal history of a fourth degree laceration during screening physical exam.
* Any other medical condition that the investigators feel would compromise the study.
* Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. bacterial vaginosis, herpes genitalis, candida).
* Stage III or IV pelvic organ prolapse.
* History of any female sexual disorder.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Microscopic evaluation for vaginal epithelial thickness | 4-5 weeks after the last treatment
  The vaginal epithelial thickness will be measured in micrometers. Then the difference in vaginal epithelial thickness between the biopsy obtained before and after the start of laser treatment will be calculated, considering a 20% increase as significant.
Microscopic evaluation of number of papillae | 4-5 weeks after the last treatment
  The number of papillae in bioptic samples will be analyzed with Hematoxylin- Eosin and Trichrome staining.
Microscopic evaluation of glycogen amount | 4-5 weeks after the last treatment
  The amount of glycogen present at the epithelial level and the ratio between the number of type I collagen fibers and type III will be evaluated with PAS reaction for glycogen.
Microscopic evaluation of number and size of the vessels | 4-5 weeks after the last treatment
  The number and size of the vessels present in the subepithelial layer will be evaluated using immunohistochemistry for CD34, a vessel marker.

SECONDARY OUTCOMES:
Validated questionnaires VHI | 4-5 weeks after the last treatment
  Vaginal Health Index (VHI) for evaluation of vaginal atrophy severity that is composed by the sum of 6 fields (min score 1 max score 5). The least score (6) is the worst; the maximum score (30) is the best.
Validated questionnaires FSFI | 4-5 weeks after the last treatment
  Female Sexual Function Index (FSFI) questionnaire which will assess female sexual function that is composed of 19 fields. The minimum score is 2 in the worst situation; maximum score is 36 in the best situation
Validated questionnaires UDI-6 | 4-5 weeks after the last treatment
  Urinary Distress Inventory-6 (UDI-6) is a 6 fields questionnaires on voiding function. The minimum score is 0 in absence of symptoms; 18 is the maximum score in the worst situation.
Validated questionnaires ICIQ-UI | 4-5 weeks after the last treatment
  International Consultation on Incontinence Questionnaire - Urinary Incontinence (ICIQ-UI) which will evaluate the extent of urinary symptoms. It is divided into two parts: questions 1, 2 and 3 are added together and the maximum score is 22, in worst condition; a score of zero is obtained in asymptomatic patients. The last is a describing question.
Validated questionnaires LIKERT | 4-5 weeks after the last treatment
  5-point Likert scale is made to assess the impact of GSM symptoms on quality of life (QoL). It is a descriptive question.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Salvatore, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cagnacci A, Xholli A, Sclauzero M, Venier M, Palma F, Gambacciani M; writing group of the ANGEL study. Vaginal atrophy across the menopausal age: results from the ANGEL study. Climacteric. 2019 Feb;22(1):85-89. doi: 10.1080/13697137.2018.1529748. Epub 2019 Jan 2. PMID 30601037
- [Background] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Salvatore S, Nappi RE, Zerbinati N, Calligaro A, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. A 12-week treatment with fractional CO2 laser for vulvovaginal atrophy: a pilot study. Climacteric. 2014 Aug;17(4):363-9. doi: 10.3109/13697137.2014.899347. Epub 2014 Jun 5. PMID 24605832
- [Derived] Casiraghi A, Calligaro A, Zerbinati N, Doglioli M, Ruffolo AF, Candiani M, Salvatore S. Long-term clinical and histological safety and efficacy of the CO2 laser for treatment of genitourinary syndrome of menopause: an original study. Climacteric. 2023 Dec;26(6):605-612. doi: 10.1080/13697137.2023.2246886. Epub 2023 Aug 31. PMID 37650754

DOCUMENTS (1):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04868812/Prot_000.pdf